CLINICAL TRIAL: NCT04771832
Title: Enhanced Recovery After Surgery (ERAS) Protocol is a Safe and Effective Approach in Patients With Gastrointestinal Fistulas Undergoing Reconstruction: Results From a Prospective Study.
Brief Title: ERAS in Gastrointerstinal Fistulas.
Status: Completed | Type: Observational
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Unit, Stanley Dudrick's Memorial Hospital
Other Study IDs: ERASGI
Record Dates: First submitted 2021-02-21; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Fistula; Surgery Site Fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERAS: Perioperative care with Enhanced Recovery After Surgery (ERAS) protocol
  Interventions: Procedure: ERAS

INTERVENTIONS:
Procedure: ERAS — Enhanced Recovery After Surgery (ERAS) protocol is an evidence-based multimodal perioperative protocol focused on stress reduction and the promotion of a return to function

SUMMARY:
An enterocutaneous fistula (ECF) poses a major surgical problem. The definitive surgical repair of persistent fistulas remains a surgical challenge with a high rate of re-fistulation and mortality, and the reasons for that is not the surgical technique alone. Enhanced Recovery after Surgery (ERAS®) is an evidence-based multimodal perioperative protocol proven to reduce postoperative complications. The aim of the study was to assess the clinical value of ERAS protocol in surgical patients with ECF.

DETAILED DESCRIPTION:
ERAS protocol was used in all patients scheduled for surgery for ECF at the Stanley Dudrick's Memorial Hospital in Skawina between 2011 and 2020. A multidisciplinary team (MDT) was in charge of the program and performed annual audits. A consecutive series of 100 ECF patients (44 F, 56 M, mean age 54.1) was evaluated. Postoperative complications rate, readmission rate, length of hospital stay, prevalence of postoperative nausea and vomiting were assessed.

ELIGIBILITY:
Inclusion Criteria:

* surgery for gastrointestinal fistula

Exclusion Criteria:

* conservative treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients scheduled for fistula surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | up to 24 weeks
  Any surgical complications
length of hospital stay | up to 24 weeks
  duration of hospitalization
postoperative nausea and vomiting | up to 24 weeks
  prevalence of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No
No sharing

REFERENCES:
- [Derived] Klek S, Salowka J, Choruz R, Cegielny T, Welanyk J, Wilczek M, Szczepanek K, Pisarska-Adamczyk M, Pedziwiatr M. Enhanced Recovery after Surgery (ERAS) Protocol Is a Safe and Effective Approach in Patients with Gastrointestinal Fistulas Undergoing Reconstruction: Results from a Prospective Study. Nutrients. 2021 Jun 7;13(6):1953. doi: 10.3390/nu13061953. PMID 34200140